CLINICAL TRIAL: NCT03767673
Title: Examination of the Cardiorespiratory Performance Capacity and Pulmonary Microbiome in Patients Following Surgical Repair of Esophageal Atresia
Brief Title: Cardiorespiratory Performance and Pulmonary Microbiome in Patients After Repair of Esophageal Atresia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1.1
Record Dates: First submitted 2018-07-19; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Esophageal Atresia
MeSH Terms: conditions — Esophageal Atresia | interventions — Aging

STUDY DESIGN:
Masking Description: Control group: Age and sex matched healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients after esophageal atresia (Experimental): Patients older than 12 years following surgical repair of congenital esophageal atresia will be included after written informed consent. Patients will be subjected to spirometry to determine their age, weight (determined by Kilogram (kg) on a medical weight scale) and Vital Capacity before (initial Spirometry) and after (final Spirometry) exercise performance testing. Bicycle ergospirometer will be applied to determine the Maximum Oxygen Uptake and the Maximum Performance. Thereafter deep induced sputum will be harvested for measurements of the pulmonary microbiome (Pulmonary Microbiome 16S rDNA profiling).
  Interventions: Diagnostic Test: Initial Spirometry; Diagnostic Test: Final Spirometry; Diagnostic Test: Pulmonary microbiome (16S rDNA profiling); Diagnostic Test: Maximum oxygen uptake; Diagnostic Test: Maximum performance; Diagnostic Test: weight; Other: age
- Control group (Active Comparator): Age and sex matched adolescents will be recruited as control group and will be included after written informed consent. Adolescents will be subjected to spirometry to determine their age, weight (determined by Kilogram on a medical weight scale) and Vital Capacity before (initial Spirometry) and after (final Spirometry) exercise performance testing. Bicycle ergospirometer will be applied to determine the Maximum Oxygen Uptake and the Maximum Performance. Thereafter deep induced sputum will be harvested for measurements of the pulmonary microbiome (Pulmonary Microbiome 16S rDNA profiling).
  Interventions: Diagnostic Test: Initial Spirometry; Diagnostic Test: Final Spirometry; Diagnostic Test: Pulmonary microbiome (16S rDNA profiling); Diagnostic Test: Maximum oxygen uptake; Diagnostic Test: Maximum performance; Diagnostic Test: weight; Other: age

INTERVENTIONS:
Diagnostic Test: Initial Spirometry — Determination of Vital Capacity by spirometry before (within 30 minutes) spiroergometry. Measurements will be performed in both groups.
Diagnostic Test: Final Spirometry — Determination of Vital Capacity by spirometry after (within 30 minutes) spiroergometry. Measurements will be performed in both groups.
Diagnostic Test: Pulmonary microbiome (16S rDNA profiling) — Harvesting of deep induced sputum and determination of the airway microbiome by 16S ribosomal RNA (rRNA) pyrosequencing. Evaluation of alpha and beta diversity and relative bacterial abundance at the genus level. Measurements will be performed in both groups (samples will be harvested within 30 minutes after spiroergometry).
Diagnostic Test: Maximum oxygen uptake — Determination of the maximum oxygen uptake (ml/kg/min) corrected for gender, age and body weight by bicycle spiroergometry. Measurements will be performed in both groups.
Diagnostic Test: Maximum performance — Determination of the maximum performance (W/kg) corrected for body weight by bicycle spiroergometry. Measurements will be performed in both groups.
Diagnostic Test: weight — Determined by Kilogram on a medical weight scale
Other: age — Determination of age by patient's Report and past medical history

SUMMARY:
The majority of the clinical research on esophageal atresia focuses on the upper gastrointestinal tract. However, the trachea and the lung are also affected in many of these children, so that a lifelong pulmonary impairment may result. The importance of respiratory function in the context of follow-up of these patients has therefore been increasingly recognized in recent years. Scientific work has shown significantly, that patients following esophageal atresia repair develop respiratory symptoms more frequently than the normal population. Mild impairment of the pulmonary function in adolescence and adulthood was demonstrated in some studies, but to date, there is no exact idea about the relationship between early childhood disease progression and later pulmonary impairment. Only a few scientific papers have dealt with the effect of impaired pulmonary function on the physical capacity of these adolescents and adults. Most of these studies show small case numbers, inconclusive stress tests, and divergent results.

The aim of this prospective study is to investigate the cardiopulmonary performance capacity and the pulmonary microbiome of adolescent and adult patients with corrected esophageal atresia and to compare the results with a control group. Another focus of the investigators is on the composition of the pulmonary microbiome of the participants. Changes of the pulmonary microbiome and the influence on the cardio-pulmonary performance capacity have not yet been investigated. Furthermore, it should be investigated whether the treatment measures and a complicated disease course in the neonatal period have long-term effects on lung function, exercise capacity and composition of the microbiome in the lungs.

ELIGIBILITY:
Inclusion Criteria:

* Age from 12 years
* Status post surgical correction of esophageal atresia with and without fistula
* Granted consent

Exclusion Criteria:

* Acute infections within the last 14 days
* Other associated serious malformations
* Acute, temporary respiratory complaints (cough, allergies etc.)
* Physical and mental illnesses or disabilities that do not allow the examination to be carried out
* non-granted consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-04-06 (Estimated); Study Completion 2019-09-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary microbiome (16S rDNA profiling) - Alpha diversity | 1 year
  Determination of alpha diversity (Chao1 Test) at the genus level of deep induced Sputum by 16S rDNA profiling. Comparison of Alpha diversity (Chao1 Analysis) between patients after repair of esophageal atresia and age and sex matched healthy controls.
Pulmonary microbiome (16S rDNA profiling) - Beta diversity | 1 year
  Determination of beta diversity (unweighted UniFrac test) at the genus level of deep induced Sputum by 16S rDNA profiling. Comparison of beta-diversity (Unweighted UniFrac Analysis) between patients after repair of esophageal atresia and age and sex matched healthy controls.
Pulmonary microbiome (16S rDNA profiling) - relative bacterial abundance | 1 year
  Determination of relative bacterial abundance (in per Cent) at the genus level of deep induced Sputum by 16S rDNA profiling. Comparison of relative bacterial abundance (Mann-Whitney-U-Test) between patients after repair of esophageal atresia and age and sex matched healthy controls.

SECONDARY OUTCOMES:
Maximum oxygen uptake (ergospirometer) | 1 year
  Maximum oxygen uptake (corrected for age, gender and body weight ) as determined by bicycle ergospirometer. Comparison of parameters between patients after repair of esophageal atresia and age and sex matched healthy controls.
Maximum Performance (ergospirometer) | 1 year
  Maximum performance as determined by bicycle ergospirometer. Comparison of parameters between patients after repair of esophageal atresia and age and sex matched healthy controls.
Vital capacity (spirometry) | 1 year
  Vital capacity as determined by spirometry. Comparison of parameters between patients after repair of esophageal atresia and age and sex matched healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Windhaber, MD, Study Director — Department of Paediatric and Adolescent Surgery, Medical University of Graz, Austria; Holger Till, MD, Study Chair — Department of Paediatric and Adolescent Surgery, Medical University of Graz, Austria; Christoph Arneitz, MD, Principal Investigator — Department of Paediatric and Adolescent Surgery, Medical University of Graz, Austria
Locations (1):
- Medical University of Graz, Graz, Austria